CLINICAL TRIAL: NCT01796626
Title: Clinical Evaluation of M22 ResurFX 1565nm Module
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-M22-ResurFX-12-01
Record Dates: First submitted 2013-02-17; First posted 2013-02-22 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Wrinkles; Striae
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wrinkle treatment (Experimental): Wrinkle treatment with ResurFX 1565nm module
  Interventions: Device: M22 ResurFX module
- Striae treatment (Experimental): Striae treatment with the REsurFX 1565nm module
  Interventions: Device: M22 ResurFX module

INTERVENTIONS:
Device: M22 ResurFX module — The system delivers pulsed near Infra-Red (NIR) laser light with a nominal wavelength of 1565 nm and has a unique treatment handpiece with epidermal cooling. The clinician is able to control the settings of energy, µBeams density, scan size, and shape option from the user interface (LCD GUI) display on the main M22 console.

SUMMARY:
At least thirty (30) subjects, Fitzpatrick-Goldman Skin Type I-IV will be enrolled in 2 clinical sites; each clinic will enroll at least 15 subjects.

Subjects should present visible wrinkles and/or striae requiring treatment.

Hypothesis: The M22 ResurFX 1565nm module will improve the appearance of the wrinkles by at least 2 grades on the Fitzpatrick-Goldman Wrinkle and Elastosis Score, and striae by at least 50% using VAS as compared to baseline, for at least 75% of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand and provide written Informed Consent;
* Healthy adult, male or female, 25-55 years of age with Fitzpatrick-Goldman skin type I-IV;
* Having suitable areas of treatment of facial areas to be treated with wrinkles Fitzpatrick-Goldman Wrinkle and Elastosis Score of 3-6 or striae alba present for more than 1 year;
* Able and willing to comply with the treatment/follow-up schedule and requirements;
* Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

Any of the following will exclude the subject from the study: skin type V-VI

1. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding;
2. History of post inflammatory hyperpigmentation
3. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study;
4. Use of photosensitive medication for which light exposure is contraindicated.
5. Use of oral isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study. Note: skin must regain its normal degree of moisture prior to treatment;
6. Prior treatment, such as chemical peel (especially phenol based) or dermabrasion, in treated area within 3 months of initial treatment or during the course of the study;
7. Prior skin treatment with non-ablative laser or other devices in treated area within 6 months of initial treatment or during the course of the study;
8. Prior use of collagen, fat injections or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 12 months of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants;
9. Prior use of Botox in treatment area within 6 months;
10. Prior ablative resurfacing procedure or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study;
11. Any other surgery in treated area within 9 months of initial treatment or during the course of the study;
12. History of keloid or any other type of hypertrophic scar formation or poor wound healing in a previously injured skin area;
13. Showing symptoms of hormonal disorders, as per the Investigator's discretion (such as Melasma, Chloasma);
14. Concurrent inflammatory skin conditions, including, but not limited to, rosacea of any severity;
15. Open laceration or abrasion of any sort on area to be treated during the course of treatment;
16. Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment;
17. Multiple dysplastic nevi in area to be treated;
18. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to treatment (as per the patient's physician discretion);
19. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications;
20. Having any form of active cancer at the time of enrollment and during the course of the study or history or skin cancer;
21. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process; Participation in a study of another device or drug within 3 month prior to study enrollment or during this study, and as per the Investigator's discretion, as long as not contradictory to any of the above criteria;
22. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
23. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Improvement | 3 months following 3rd treatment
  Investigator subjective evaluation of the extent of wrinkles improvement at the 3 month follow-up visit as assessed by Fitzpatrick-Goldman Wrinkle Class / Elastosis Score classification, striae improvement will be assessed using VAS.

SECONDARY OUTCOMES:
Improvement | 1 and 6 months following 3rd treatment
  Investigator subjective evaluation of the extent of wrinkles/striae improvement by the investigator at 1 and 6 month follow-up visits as assessed by Fitzpatrick-Goldman Wrinkle Class / Elastosis Score classification, striae improvement will be assessed using VAS.
Blinded improvement | 1 year following study initiation
  Blinded evaluation of wrinkles/striae skin improvement at the 1, 3 and 6 months follow-up as compared to baseline using photographs may be performed at the end of the study.
Skin response | Following treatment #1, 2 and 3
  Investigator subjective evaluation of skin response following each treatment defined as severity of response and the time it took for it subside
Downtime | Following treatment #1, 2 and 3
  Downtime defined as the period of time following the procedure during which the subject felt uncomfortable, unwilling or unable to go out in public due to edema and erythema
Improvement by subject | 1, 3 and 6 months follow up
  Subject subjective opinion of improvement and satisfaction with the treatment based on a 5 point scale
Comfort | Following treatment #1, 2 and 3
  Subject subjective assessment of pain and discomfort associated with treatments using a 10 point VAS scale
Biopsies | 1, 3 and 6 months follow up
  Histological analysis of tissue samples with different staining for analysis of changes following treatment
Adverse Events | Following treatment #1, 2 and 3 and all follow up visits
  Any adverse events associated with various setting used during the treatment and follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — DCLA; Arielle NB Kauvar, MD, Study Director — New York Laser & Skin Care
Locations (2):
- United States (2):
  - DCLA, San Diego, California
  - New York Laser & Skin Care, New York, New York